CLINICAL TRIAL: NCT04476342
Title: Integration of Minimal Invasive Cardiopulmonary Bypass System and the Research of Its Blood Compatibility
Acronym: IMICPBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-044
Record Dates: First submitted 2020-06-28; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-06

CONDITIONS: Cardiopulmonary Bypass; Cardiac Surgery
Keywords: cardiopulmonary bypass; minimal invasive; cardiac surgery; blood compatibility
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MICPB group (Experimental): The experimental group is minimal invasive cardiopulmonary bypass (MICPB) group, with built-in micro-thrombotic oxygenator and mini cardioplegia (MP) formula (15ML15% KCl+10ml compound potassium, calcium and magnesium +25ml normal saline).
  Interventions: Device: minimal invasive cardiopulmonary bypass (MICPB) system
- CCPB group (No Intervention): The control group was conventional cardiopulmonary bypass (CCPB) group, using ordinary oxygenator, microemboli filter, and 4:1 cardioplegia solution.

INTERVENTIONS:
Device: minimal invasive cardiopulmonary bypass (MICPB) system — The experimental group was MICPB group, with built-in micro-thrombotic oxygenator and MP formula (15mL 15%KCl+10ml compound potassium, calcium and magnesium +25ml normal saline)
  Arms: MICPB group

SUMMARY:
Research objective:

(1) To develop a minimally invasive extracorporeal circulation integrated system, and to form a new product package, the package of the system should include the extracorporeal circulation off-set supplies for a routine heart operation.(2) To explore the influence of integrated minimally invasive extracorporeal circulation system on the recent clinical outcome of patients.(3) To explore the influence of integrated minimally invasive extracorporeal circulation system on blood dilution of patients.(4) To explore the influence of integrated minimally invasive extracorporeal circulation system on inflammatory response in patients.

1) Clinical research methods: A prospective, single-blind, randomized controlled study was designed. 80 patients should be included.Clinical study grouping: The control group was conventional cardiopulmonary bypass (CCPB) group, which was equipped with ordinary oxygenator, microemboli filter and 4:1 cardioplegia solution.The experimental group was minimal invasive cardiopulmonary bypass (MICPB) group, with built-in micro-thrombotic oxygenator and mini cardioplegia (MP) formula (15ML15% potassium chloride (KCl)+10ml compound potassium, calcium and magnesium +25ml normal saline).

Research method:

A: Before, in, and after cardiopulmonary bypass (CPB) blood collection, Hemoglobin (Hb), hematokrit (Hct), and blood lactate values of the two groups of patients were measured and analyzed statistically.B: Blood transfusion volume, urine volume and ultrafiltration volume were collected during CPB in the two groups of patients, and the data of the two groups were statistically analyzed.To investigate the effects of integrated minimally invasive extracorporeal circulation system on inflammatory response indicators white blood cell count (WBC),C-reactive protein (CRP), interleukin-6(IL-6), tumor necrosis factor-a (TNF-a) and C3a in patients before (T0), CPB (T1) and 2 hours(H) after CPB (T2), blood samples were collected from the two groups, centrifugated, superfluid was taken, and stored at -80℃.The concentrations of CRP, IL-6, TNF-a and C3a were determined by ELISA.Statistical analysis was performed.WBC was measured in blood routine.(3) To investigate the influence of integrated minimally invasive extracorporeal circulation system on the recent clinical outcome of patients. The mechanical ventilation time, ICU time, length of hospital stay, and in-hospital mortality of patients in the two groups were statistically analyzed.

DETAILED DESCRIPTION:
Research objective:

(1) To develop a minimally invasive extracorporeal circulation integrated system, and to form a new product package, the package of the system should include the extracorporeal circulation off-set supplies for a routine heart operation.(2) To explore the influence of integrated minimally invasive extracorporeal circulation system on the recent clinical outcome of patients.(3) To explore the influence of integrated minimally invasive extracorporeal circulation system on blood dilution of patients.(4) To explore the influence of integrated minimally invasive extracorporeal circulation system on inflammatory response in patients.

Research and development of integrated minimally invasive extracorporeal circulation system

(1) Appropriate CPB tubes should be determined according to clinical needs. Adopt 3/8 inch vein tubes and elevate the position of blood storage tank to reduce the length of the tubes and precharge.The piping jacket shall include the main pump pipe, the infusion pipe, the platform package (static and static vessels), the left and right core suction pipe, and the negative pressure suction pipe.The total precharge should be kept at about 800ml (284ml static precharge of the self-equipped micro-plug oxygenator, and about 500ml precharge of the pipeline and stopping liquid perfusion system).(2) Cooperate with integrated membrane oxygenator manufacturers in the design of pipelines to form a wrapper that integrates membrane oxygenator and pipeline.Among them, oxygenator and pipeline should be well connected in the sheath.

Clinical research methods:

A prospective, single-blind, randomized controlled study was designed. 80 patients should be included.Clinical study grouping: The control group was CCPB group, which was equipped with ordinary oxygenator, microemboli filter and 4:1 cardioplegia solution.The experimental group was MICPB group, with built-in micro-thrombotic oxygenator and MP formula (15ML15% KCl+10ml compound potassium, calcium and magnesium +25ml normal saline).

Research method:

A: Before, in, and after CPB blood collection, Hb, Hct, and blood lactate values of the two groups of patients were measured and analyzed statistically.B: Blood transfusion volume, urine volume and ultrafiltration volume were collected during CPB in the two groups of patients, and the data of the two groups were statistically analyzed.To investigate the effects of integrated minimally invasive extracorporeal circulation system on inflammatory response indicators WBC, CRP, IL-6, TNF- and C3a in patients before (T0), CPB (T1) and 2 hours after CPB (T2), blood samples were collected from the two groups, centrifugated, superfluid was taken, and stored at -80℃.The concentrations of CRP, IL-6, TNF- and C3a were determined by ELISA.Statistical analysis was performed.WBC was measured in blood routine.(3) To investigate the influence of integrated minimally invasive extracorporeal circulation system on the recent clinical outcome of patients. The mechanical ventilation time, ICU time, length of hospital stay, and in-hospital mortality of patients in the two groups were statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient weight ≤60kg;
* Age ≥18 years old;
* The patient underwent cardiac arrest surgery.

Exclusion Criteria:

* Heart transplant patients;
* Emergency cardiac surgery patients;
* Patients who had been assisted by extracorporeal membrane oxygenator (ECMO) or assisted by left heart before operation
* Left ventricular ejection fraction (LVEF) < 30%;
* Patients with coagulation dysfunction before surgery;
* Patients with preoperative hepatic and renal insufficiency;
* Recent cerebrovascular accident patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood transfusion volume | through surgery completion, an average of 5 hours
  Blood transfusion volume during cardiac surgery

SECONDARY OUTCOMES:
ICU duration | Duration of ICU stay, an average of 3 days
  Duration of ICU Stay

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No